CLINICAL TRIAL: NCT06207838
Title: Transition of T1DM Patients Aged Over 65 Years Into AHCL (780G) Insulin Pump: the Impact on Glucose Patterns, Quality of Life Physical & Cognitive Measures, as Well as Vascular Status
Brief Title: Transition of T1DM Patients Aged Over 65 Years Into AHCL (780G) Insulin Pump
Acronym: 780G65+
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Jagiellonian University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Tomasz Klupa, Prof. Tomasz Klupa, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1072.61201.5.2023
Record Dates: First submitted 2023-05-16; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Type 1
Keywords: AHCL; Insulin pump therapy; Multiple daily injection; QoL
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: The trial is a two-centers, randomized controlled, parallel group study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Actual therapy (No Intervention): The patient continues Multiple Daily Injection/Insulin Pump Therapy with or without CGM use as per routine procedures
- Advanced Hybrid Cloosed Loop System (Experimental): The patients will be switched to MiniMed 780G advanced hybrid cloosed loop system/ AHCL system
  Interventions: Device: MiniMed 780G system

INTERVENTIONS:
Device: MiniMed 780G system — The MiniMed™ 780G system automatically adjust insulin delivery to patient needs for an easier way to stabilise glucose levels. It features an advance level of automation for diabetes management, known as SmartGuard™ technology. If patient glucose levels are trending high, it gives patient more insulin. Technology is CE marked.
  Arms: Advanced Hybrid Cloosed Loop System

SUMMARY:
Older people with diabetes have a higher risk for cognitive impairment and for physical disability whether this may be effected by an improvement in glucose indices is unknown. Thus, the aim of this study is to assess the efficacy of AHCL in people with type 1 diabetes in improving glucose indices, quality of life and physical capacity indices

DETAILED DESCRIPTION:
Recent advances in insulin pumps, continuous glucose monitoring (CGM) devices, and control algorithms have resulted in an acceleration of progress in the development of the automated systems of insulin delivery including advanced hybrid closed loop (HCL) insulin pumps. The results of the AHCL insulin pump based studies published so far are very encouraging, including that Medtronic-sponsored study performed at our center "Transition of CSII/CGM naïve patients directly into AHCL (780G) insulin pump: the impact on glucose patterns and quality of life measures" (1-6). Unfortunately there is little data concerning the usage of AHCL systems in older patients. The management of these individuals is particularly challenging as older adults with type 1 diabetes are especially vulnerable to hypoglycaemia. The recent ADA/EASD consensus underlines that the use of advanced technologies in older individuals is useful and should not be discontinued or a priori excluded because of the older age (7). Since the AHCL systems are very effective in hypoglycemia prevention they could be considered the treatment of choice in older patients with T1DM. The open question is how effectively would older individuals adopt this advanced technology, how would they accept it, and if the simplicity in terms of everyday usage of AHCL versus less advanced technologies would be appreciated by older individuals with T1DM. Older people with diabetes have a higher risk for cognitive impairment and for physical disability whether this may be effected by an improvement in glucose indices is unknown. Thus, the aim of this study is to assess the efficacy of AHCL in people with type 1 diabetes in improving glucose indices, quality of life and physical capacity indices

ELIGIBILITY:
Inclusion Criteria:

1. Age over 65 years
2. T1DM
3. Willing to participate in a study for the specified duration
4. Willing to perform ≥ 4 finger stick blood glucose measurements daily
5. Willing to wear the system continuously throughout the study
6. Glycosylated hemoglobin (A1C) value less than 10.0% at time of screening visit
7. Treated with MDI/CSII (with exclusion of 780G)
8. Willing to perform at least 4 BGM/day, when on MDI/CSII
9. Lack of advanced complications of diabetes, eGFR>30

Exclusion Criteria:

1. Severe concurrent illness
2. Laboratory abnormalities, or medications that might affect study participation,
3. Severe renal impairment (eGFR<30)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2024-09-07 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Between group difference in the percentage of time spent within range with sensor glucose (SG) between 70-180 mg/dL (TIR) (3.9-10.0 mmol/L). | Month 12
  Between group difference in the percentage of time spent within range with sensor glucose (SG) between 70-180 mg/dL (TIR) (3.9-10.0 mmol/L).

SECONDARY OUTCOMES:
Between groups difference in the percentage of participants achieving TIR >70% | Month 12
  Between groups difference in the percentage of participants achieving TIR >70%
Between group difference in the percentage of time spent in hyperglycemic range with SG > 250 mg/dL (13.9 mmol/L) | Month 12
  Between group difference in the percentage of time spent with SG > 250 mg/dL (13.9 mmol/L)
Between group difference in the percentage of time spent in hyperglycemic range with SG > 180 mg/dL (10.0 mmol/L) | Month 12
  Between group difference in the percentage of time spent with SG > 180 mg/dL (10.0 mmol/L)
Between group difference in the percentage of time spent in hypoglycemic range with SG < 54 mg/dL (3.0 mmol/L) | Month 12
  Between group difference in the percentage of time spent in hypoglycemic range with SG < 54 mg/dL (3.0 mmol/L)
Between group difference in the percentage of time spent in hyperglycemic range in hypoglycemic range with SG < 70 mg/dL (3.9 mmol/L) | Month 12
  Between group difference in the percentage of time spent in hyperglycemic range in hypoglycemic range with SG < 70 mg/dL (3.9 mmol/L)
QoL group difference using: The World Health Organisation- Five Well-Being Index (WHO-5) | Month 12
  QoL group difference (WHO-5): Final score: 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
Differences in baseline vs end of the study in vascular status as measured with LDF: Laser Doppler Flowmetry | Month 12
  Differences in baseline vs end of the study in vascular status as measured with LDF: Laser Doppler Flowmetry
Differences in baseline vs end of the study in vascular status as measured with FMD: Flow-Mediated Dilatation | Month 12
  Differences in baseline vs end of the study in vascular status as measured with FMD: Flow-Mediated Dilatation
Differences in baseline vs end of the study in vascular status as measured with IMT-Intima-media thickness | Month 12
  Differences in baseline vs end of the study in vascular status as measured with IMT-Intima-media thickness,
Difference in physical capacity indices listed in screening visit: 6 Minute Walk Test | Month 12
  Difference in physical capacity indices listed in screening visit: 6 Minute Walk Test (units distance in meters, higher value mean a better outcome)
Difference in physical capacity indices listed in screening visit: Fried Scale | Month 12
  Difference in physical capacity indices listed in screening visit: Fried Scale (higher scores mean a worse outcome, score >3 frail present)
Difference in physical capacity indices listed in screening visit: Berg Balance Scale | Month 12
  Difference in physical capacity indices listed in screening visit: Berg Balance Scale (higher score mean a better outcome)
Difference in physical capacity indices listed in screening visit: Four Square Step | Month 12
  Difference in physical capacity indices listed in screening visit:Four Square Step (units time, shorter time means better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Klupa, Prof., Principal Investigator — Jagiellonian University
Locations (1):
- Hospital University; Jagiellonian University Medical College, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/38/NCT06207838/Prot_000.pdf